CLINICAL TRIAL: NCT05701527
Title: A Phase 1A/B Study To Evaluate The Safety And Tolerability Of EBC-129 As A Single Agent And In Combination With Pembrolizumab In Advanced Solid Tumours
Brief Title: A Study of EBC-129 in Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EDDC (Experimental Drug Development Centre), A*STAR Research Entities (Other Government)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBC-129-01
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumours
Keywords: Advanced solid tumours; Antibody drug conjugates (ADCs); Recommended phase-2 dose (RP2D); Monomethyl auristatin E (MMAE); N-glycosylated CEACAM5/6
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A-Cohort 1 (Experimental): Patients will be administered Dose 1 of EBC-129 as a monotherapy.
  Interventions: Drug: EBC-129
- Part A-Cohort 2 (Experimental): Patients will be administered Dose 2 of EBC-129 as a monotherapy.
  Interventions: Drug: EBC-129
- Part A-Cohort 3 (Experimental): Patients will be administered Dose 3 of EBC-129 as a monotherapy.
  Interventions: Drug: EBC-129
- Part A-Cohort 4 (Experimental): Patients will be administered Dose 4 of EBC-129 as a monotherapy.
  Interventions: Drug: EBC-129
- Part A-Cohort 5 (Experimental): Patients will be administered Dose 5 of EBC-129 as a monotherapy.
  Interventions: Drug: EBC-129
- Part B (Experimental): Patients will be administered three different dose levels of EBC-129 in combination with a fixed dose of pembrolizumab.
  Interventions: Drug: EBC-129; Drug: Pembrolizumab
- Part C (Experimental): Patients will be administered the highest dose of EBC-129 as a monotherapy at the RP2D determined in Part A of the study.
  Interventions: Drug: EBC-129
- Part D: EBC-129 (Experimental): Patients will be administered EBC-129 as a monotherapy as per two-dose or three-dose per cycle regimen.
  Interventions: Drug: EBC-129

INTERVENTIONS:
Drug: EBC-129 — EBC-129 will be administered on Day 1 of each 21-Day cycle (Parts A, B, and C), and two doses starting from Day 1 for 21-day cycle and three doses starting from Day 1 for 28-day cycle (Part D) via a 30-120-minute intravenous (IV) fusion.
Drug: Pembrolizumab — Pembrolizumab will be administered at the dose of 200 mg IV every 21 days.
  Arms: Part B

SUMMARY:
This study will assess the safety and tolerability of EBC-129 as a single agent and in combination with pembrolizumab in patients with advanced solid tumours

DETAILED DESCRIPTION:
This study is a prospective, open label study which is divided into 4 parts.

Part A will be dose escalation segment to identify the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of EBC-129 monotherapy.

Part B will be dose escalation segment to identify the MTD and RP2D of EBC-129 in combination with pembrolizumab.

Part C (dose expansion cohort) will be performed in an expanded cohort of patients with advanced solid malignancies at the RP2D of EBC-129 as a monotherapy identified in the dose escalation segment, Part A.

Part D (Dose Fractionation Cohort) will be performed in patients with advanced solid malignancies with cancer indications that have shown preliminary clinical activity in Part C.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years (US) or ≥21 years (Singapore) old
2. Body weight within ≥40 kg - ≤100 kg during Parts A and B, and ≤120 kg during all other parts of the study
3. Demonstrated progression of a locally advanced unresectable or metastatic solid tumour with no alternative standard-of-care therapeutic option with a proven clinical benefit, or are intolerant to these therapies
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2 for Part A and 0-1 for Parts B, C and D
5. Hepatic function and adequate renal function, as per protocol standard
6. Adequate bone marrow function as per protocol standard

Exclusion Criteria:

1. Unable or not willing to provide tumour tissue sample (from archival tissue or de-novo biopsy) unless if there is a significant risk for the patient to undergo biopsy
2. Has received investigational or anti-cancer therapy within 4 weeks (28 days) prior to starting study drug
3. Is receiving any concomitant anti-cancer therapy
4. Known severe hypersensitivity to E coli-derived products or filgrastim or peg-filgrastim and have significant allergies to such biological products
5. Has clinically active brain metastases
6. Has received prior radiation therapy
7. Has received prophylactic administration of haematopoietic colony stimulating factors within 4 weeks (28 days) prior to starting study drug
8. Patients concurrently using any strong P-glycoprotein (P-gp) inducers/inhibitors or strong cytochrome P3A (CYP3A) inhibitors within 14 days prior to the first dose of study drug or patients that use restricted or prohibited medications listed in the concomitant and other treatments section of the protocol
9. Pregnancy or breast feeding
10. For patients receiving pembrolizumab:

    1. Has an active autoimmune disease that has required systemic treatment in the past 2 years
    2. Patients who, according to the currently approved Keytruda (pembrolizumab) US package insert (USPI)/summary of product characteristics, had an immune-related adverse event (irAE) for which permanent discontinuation is mandated (any Grade 4 event and Grade 3 events of pneumonitis, hepatitis, and nephritis). Also, patients without formal contraindication due to previous irAE with any immune checkpoint inhibitor (approved or investigational) are not eligible if the AE has not resolved to grade 1 or better and/or still requires steroids (>10 mg of prednisone equivalent per day) for ongoing management.
    3. Patients with a history of pneumonitis/interstitial lung disease, patients who received live vaccines within 30 days of enrolment, and patients who discontinued prior immune checkpoint inhibitors due to Grade 2 myocarditis are excluded from enrolment into pembrolizumab-containing cohorts
11. Has had a major surgical procedure within 4 weeks (28 days) from starting the study drug
12. Patients with active or chronic corneal disorders, with other active ocular conditions requiring ongoing therapy or with any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy
13. Active infection including HIV, Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Part A, Part B, Part C and Part D- Number of patients with serious adverse events (SAEs) and treatment emergent adverse events (TEAEs) | From pre-screening (≥28 days from planned date of treatment i.e. Day 1) until end of study (EOS i.e., 30 days from last dose). Approximately 2 years
Part A, Part B and Part D- Determination of Maximum tolerated dose (MTD) | Approximately 2 years
Part A, Part B and Part D- Determination of the Recommended Phase 2 dose (RP2D) | Approximately 2 years
Part C- Objective response rate (ORR) | Day 1 through 12 cycles (each cycle is 21 days)
  The number (%) of patients with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by investigator.
Part D- ORR | Day 1 through 12 cycles (each cycle is 21 or 28 days)
  The number (%) of patients with a best overall response of CR or PR per RECIST v1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Part A and Part B- ORR | Day 1 through 12 cycles (each cycle is 21 days)
  The number (%) of patients with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by investigator.
Part A, Part B, Part C and Part D- Disease control rate (DCR) | Approximately 3.3 years
  The percentage of patients who have a best overall response (BOR) of CR or PR in the first 12 weeks or who have demonstrated standard deviation (SD) for a minimum interval of 12 weeks following the start of treatment, will be determined based on RECIST.
Part A, Part B, Part C and Part D- Duration of Response (DoR) | Approximately 3.3 years
  The time from the date of first documented response until the first date of documented progression or death in the absence of disease progression.
Part A, Part B, Part C and Part D- Time to Progression (TTP) | Approximately 3.3 years
  The time from the date of the first dose until objective tumour progression.
Part A, Part B, Part C and Part D- Progression Free Survival (PFS) | Approximately 3.3 years
  The time from the date of first dose until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anti-cancer therapy prior to progression.
Part A, Part B, Part C and Part D- Overall Survival (OS) | Approximately 3.3 years
  The time from the date of the first dose until death due to any cause.
Part A, Part B, Part C and Part D- Maximum Plasma Concentration (Cmax) of EBC-129 | Parts A, B and C: Cycle 1, 2, 3, and Cycle 4 (each cycle is 21 days); Part D: Cycle 1 (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Trough Concentration (Ctrough) of EBC-129 | Parts A, B and C: Cycle 1, 2, 3, and Cycle 4 (each cycle is 21 days); Part D: Cycle 1 (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Area under the curve (AUC) of EBC-129 | Parts A, B, and C: Cycle 1 and Cycle 2 (each cycle is 21 days); Part D: Cycle 1 (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Maximum plasma concentration at steady state (Cmax_ss) of EBC-129 | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Trough concentration at steady state (Ctrough,ss) of EBC-129 | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Area under the curve at steady state (AUC_ss) of EBC-129 | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Accumulation ratios of EBC-129 | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Time to maximum plasma concentration (Tmax) of EBC-129 | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Half-life (t1/2) of EBC-129 | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part B- Cmax of Pemrolizumab | Day 1 through 12 cycles (each cycle is 21 days)
Part B- Ctrough of Pemrolizumab | Day 1 through 12 cycles (each cycle is 21 days)
Part B- AUC of Pemrolizumab | Cycle 1 and 2 (each cycle is 21 days)
Part B- Tmax of Pemrolizumab | Day 1 through 12 cycles (each cycle is 21 days)
Part B- t1/2 of Pemrolizumab | Day 1 through 12 cycles (each cycle is 21 days)
Part A, Part B, Part C and Part D- Number of patients with detectable Anti-drug antibodies (ADAs) | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A, Part B, Part C and Part D- Number of patients with neutralising antibodies | Parts A, B, and C: Day 1 through 12 cycles (each cycle is 21 days); Part D: Day 1 through 12 cycles (each cycle is 21 or 28 days)
Part A- Comparison of tumour responses | Approximately 1.8 years
  The tumour responses (RECIST 1.1) will be compared between preselected patients and not pre-selected/not expressing the antigen when centrally assessed by immunohistochemistry (IHC).

CONTACTS AND LOCATIONS:
Overall Officials: Venkateshan Srirangam Prativadibhayankara, MD, Study Director — EDDC (Experimental Drug Development Centre), A*STAR Research Entities
Locations (5):
- United States (2):
  - University of Colorado Hospital (UCH) - University of Colorado Cancer Center (UCCC) - Neuroendocrine Tumor Center, Aurora, Colorado
  - UT MD Anderson Cancer Center, Houston, Texas
- Singapore (2):
  - National University Hospital - Medical Oncology, Singapore, South West
  - National Cancer Centre Singapore, Singapore, South West
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan